CLINICAL TRIAL: NCT02987270
Title: Evaluation of Community-based Screening and Treatment for Malaria in the KEMRI/CDC Health and Demographic Surveillance System (HDSS) in Western Kenya
Brief Title: Evaluation of Community-based Mass Screening and Treatment for Malaria in Western Kenya
Acronym: MSaT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Simon Kariuki (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Simon Kariuki, Malaria Branch Chief, Kenya Medical Research Institute
Organization: Kenya Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2380
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Malaria,Falciparum
Keywords: mass screen and treat; malaria; asymptomatic infections; transmission reduction; infectious reservoir; kenya
MeSH Terms: conditions — Malaria, Falciparum; Malaria; Asymptomatic Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mass screening and treatment (Experimental): Each member (approximately 30,000 individuals) residing within the mass screening and treatment arm were visited three times a year and tested for malaria by rapid diagnostic test; those testing positive were treated with an appropriate antimalarial- dihydroartemisinin-piperaquine was the first-line therapy. Long-lasting insecticidal net (LLIN) coverage was topped up prior to the intervention to universal coverage (one bednet for every two household participants).
  Interventions: Drug: Dihydroartemisinin-piperaquine
- Control arm (No Intervention): Members of the control arm received standard of care, which includes universal (LLIN) coverage and standard malaria case management (laboratory confirmation prior to antimalarial treatment) at the study health facilities.

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — Dihydroartemisinin-piperaquine is an antimalarial in the artemisinin-based combination therapy class of drugs. It is the Kenya Ministry of Health second-line treatment for malaria in Kenya.
  Other Names: Eurartesim
  Arms: Mass screening and treatment

SUMMARY:
This study is a cluster-randomized controlled trial to evaluate the efficacy of community-based mass screening with a malaria rapid diagnostic test, and treatment of participants with positive tests with an appropriate antimalarial for reducing malaria transmission indices.

DETAILED DESCRIPTION:
The investigators purposively selected ten health facilities in Siaya County, western Kenya based on malaria case loads. All villages whose midpoint was located within a 3 kilometer radius of each of the ten health facilities were included in the study. Contiguous villages were merged to form two clusters around each health facility. Clusters were randomly assigned to the control or intervention arm such that there was one control and one intervention cluster around each health facility. Approximately 30,000 and 60,000 people resided in intervention and control arms, respectively.

Once a year during the peak malaria transmission season in July, starting at baseline, the investigators selected a simple random sample of compounds within the study area for a cross-sectional survey to determine risk factors for malaria acquisition and parasite prevalence. Every person in each selected compound was consented into the cross-sectional survey. Community health volunteers (CHV) were trained to perform malaria rapid diagnostic tests, collect dried blood spots on filter papers, and provide treatment and referral recommendations for participants. Three times a year, in September, January, and April, for two years, CHVs visited every household in the intervention arm and tested and treated every consenting household member who was positive for malaria by rapid diagnostic test. Throughout the study period, malaria case counts from individuals located within the study clusters were recorded at each of the study health facilities. During the first two cross-sectional surveys we randomly selected 660 individuals to enter into an incidence cohort, 330 per arm. Cohort members were definitively treated for malaria at recruitment with artemether-lumefantrine, and were asked to visit a study health facility once a month for blood draws for malaria testing.

Every month, 18 households were randomly selected for entomological monitoring; 12 in the control arm, and 6 in the intervention arm. Pyrethrum spray catches were performed in each household. Live catches were performed one week in each month of the study. During live collection weeks, as many households were visited as possible, and prokopak aspirators were used to collect mosquitoes from the inner walls of houses.

Prior to the first round of mass screening and treatment and then again after the first round, 36 focus group discussions were conducted to evaluate community acceptance of community-based mass screening and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Cross sectional studies: Living within one of the study clusters, >1 month of age
* Cohort: Living within one of the study clusters, ≥1 year of age
* Passive surveillance: Living within one of the study clusters
* Entomological surveillance- household in either control or intervention arm

Exclusion Criteria:

* Cohort study- pregnant at time of recruitment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90000 (Actual)
Dates: Start 2013-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria infection | After year 1 and after year 2
  Incidence of malaria infection as determined by malaria blood smear microscopy in members of the cohort after year 1 and year 2 of mass screening and treatment

SECONDARY OUTCOMES:
Prevalence of malaria infection | After year 1 and after year 2
  Prevalence of malaria infections diagnosed by blood smear microscopy were determined during three cross-sectional studies at baseline, after year 1, and after year 2.
Incidence of clinical malaria | After year 1 and after year 2
  Incidence of clinical malaria as determined by passive surveillance in the ten study health facilities, after year 1 and after year 2.
Entomological indices of transmission | After year 1 and after year 2
  Sporozoite and oocyst rates were compared in malaria vectors captured during pyrethrum spray catches and aspirations after year 1 and after year 2.

CONTACTS AND LOCATIONS:
Overall Officials: Meghna R Desai, PhD, Principal Investigator — Centers for Disease Control and Prevention; Simon K Kariuki, PhD, Principal Investigator — Kenya Medical Research Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shuford K, Were F, Awino N, Samuels A, Ouma P, Kariuki S, Desai M, Allen DR. Community perceptions of mass screening and treatment for malaria in Siaya County, western Kenya. Malar J. 2016 Feb 6;15:71. doi: 10.1186/s12936-016-1123-y. PMID 26852227
- [Derived] Samuels AM, Odero NA, Odongo W, Otieno K, Were V, Shi YP, Sang T, Williamson J, Wiegand R, Hamel MJ, Kachur SP, Slutsker L, Lindblade KA, Kariuki SK, Desai MR. Impact of Community-Based Mass Testing and Treatment on Malaria Infection Prevalence in a High-Transmission Area of Western Kenya: A Cluster Randomized Controlled Trial. Clin Infect Dis. 2021 Jun 1;72(11):1927-1935. doi: 10.1093/cid/ciaa471. PMID 32324850